CLINICAL TRIAL: NCT01016496
Title: Rehabilitation Strategies in Children With Neuro-motor Disorders Due to the Impairment of the Central Nervous System or the Peripheral Nervous System
Brief Title: New Perspectives in the Rehabilitation of Children With Motor Disorders : the Role of the Mirror Neuron System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stefania Costi (Other)
Collaborators: University of Parma (Other); IRCCS Fondazione Stella Maris (Other)
Responsible Party: Sponsor-Investigator, Stefania Costi, technician, University of Modena and Reggio Emilia
Organization: University of Modena and Reggio Emilia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIRROR_UDGEE_09
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Hemiplegia; Cerebral Palsy
Keywords: Cerebral Palsy; Mirror neurons; hemiplegia; action observation therapy; children affected by hemiplegia as a consequence of Cerebral Palsy
MeSH Terms: conditions — Hemiplegia; Cerebral Palsy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor

ARMS (2):
- Action observation plus repetition (Experimental): Observation of actions and repetition of the same actions
  Interventions: Other: action observation therapy
- repetition only (Active Comparator): repetition of gestures
  Interventions: Other: repetition of gestures

INTERVENTIONS:
Other: action observation therapy — 15 consecutive sessions of 18 minutes, plus repetition
  Arms: Action observation plus repetition
Other: repetition of gestures — 15 consecutive session of visual games, plus repetition of gestures
  Arms: repetition only

SUMMARY:
Evidence exists that the activation of actions activates the same cortical motor areas that are involved in the performance of the observed actions. The neural substrate for this phenomena is the mirror neuron system. It is generally assumed that mirror neurons have a basic role in understanding the intentions of others and in imitation learning. There is evidence that action observation has a positive effect on rehabilitation of motor disorders after stroke. The aim of this study is to demonstrate that action observation followed by the repetition of the actions previously observed has a positive impact on rehabilitation of the upper limb in children affected by hemiplegia as a consequence of Cerebral Palsy. In particular, the purpose is to assess if mirror neurons could improve the amount, the quality and the velocity of movements and the cooperation between the two upper extremities.

ELIGIBILITY:
Inclusion Criteria:

* children with hemiplegia and
* Melbourne assessment > 50 points

Exclusion Criteria:

* inability to collaborate
* pharmacoresistant epilepsy
* inability to imitate gestures
* sensitivity disorders

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2010-05 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Melbourne Assessment of unilateral limb function | T0=baseline, Tend (week three) , T2(two months) T6months (six months after the completion of the training)

SECONDARY OUTCOMES:
Assisting Hand Assessment | T0, Tend, T2, T6
Jebsen-Taylor | T0, Tend, T2, T6
Abilhand emikids | T0, Tend, T2, T6

CONTACTS AND LOCATIONS:
Overall Officials: Rizzolatti Giacomo, Professor, Principal Investigator — University of Parma; Ferrari Adriano, Professor, Study Director — University of Modena and Reggio Emilia
Locations (3):
- Italy (3):
  - Hospital of Parma, Parma, Parma
  - IRCCS Stella Maris, Pisa, Pisa
  - Azienda Santa Maria Nuova -, Reggio Emilia, Reggio Emilia

REFERENCES:
- [Derived] Sgandurra G, Biagi L, Fogassi L, Ferrari A, Sicola E, Guzzetta A, Tosetti M, Cioni G. Reorganization of action observation and sensory-motor networks after action observation therapy in children with congenital hemiplegia: A pilot study. Dev Neurobiol. 2020 Sep;80(9-10):351-360. doi: 10.1002/dneu.22783. Epub 2020 Oct 28. PMID 32986904
- [Derived] Sgandurra G, Ferrari A, Cossu G, Guzzetta A, Biagi L, Tosetti M, Fogassi L, Cioni G. Upper limb children action-observation training (UP-CAT): a randomised controlled trial in hemiplegic cerebral palsy. BMC Neurol. 2011 Jun 28;11:80. doi: 10.1186/1471-2377-11-80. PMID 21711525